CLINICAL TRIAL: NCT00570193
Title: Photodynamic and Pharmacologic Treatment of Choroidal Neovascularization (Photodynamic Booster Study)
Brief Title: Photodynamic and Pharmacologic Treatment of CNV
Acronym: PBS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mid-Atlantic Retina Consultations, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PBS-100-388
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Choroidal Neovascularization; Macular Degeneration
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Verteporfin; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- I (Experimental): Combined treatment with verteporfin (Visudyne) and ranibizumab (Lucentis)
  Interventions: Drug: verteporfin (Visudyne)
- II (Experimental): Treatment with ranibizumab (Lucentis)
  Interventions: Drug: ranibizumab (Lucentis)

INTERVENTIONS:
Drug: verteporfin (Visudyne) — Verteporfin (Visudyne) 6 mg/m2 at 300mW/cm2 given on week O and then at week 5, given as indicated per protocol; ranibizumab (Lucentis) 0.3 mg given at week 1
  Other Names: Visudyne = verteporfin; Lucentis = ranibizumab
  Arms: I
Drug: ranibizumab (Lucentis) — ranibizumab (Lucentis) 0.3 mg on weeks 1,5,9,13,17,21,25,29,33&37 per study protocol
  Other Names: Lucentis = ranibizumab
  Arms: II

SUMMARY:
The goal of this pilot study is to validate the use of the combination of Lucentis (ranibizumab) and Visudyne (verteporfin) in the treatment of choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD) and to explore the use of a volumetric analysis of the CNV lesion to determine disease activity, response to therapy, and as a tool for determining the need for retreatment.

ELIGIBILITY:
Inclusion Criteria:

* All previously untreated CNV secondary to MD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Visual change | 18 months

SECONDARY OUTCOMES:
Frequency of treatment | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Jabbour, MD, Principal Investigator — Mid-Atlantic Retina Consultations